CLINICAL TRIAL: NCT05165433
Title: A Multicentre, Open-label, Non-randomized, Phase 1a/1b Study of NG-350A, a Tumour-selective Anti-CD40-expressing Adenoviral Vector, in Combination With Pembrolizumab in Patients With Metastatic or Advanced Epithelial Tumours
Brief Title: Study of NG-350A Plus Pembrolizumab in Metastatic or Advanced Epithelial Tumours (FORTIFY)
Acronym: FORTIFY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG-350A-02; MK-3475-C84 (Other: Merck Sharp & Dohme LLC); KEYNOTE-C84 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-03

CONDITIONS: Epithelial Tumor; Metastatic Cancer
Keywords: NG-350A; Pembrolizumab; Akamis Bio Ltd; PsiOxus; Merck
MeSH Terms: conditions — Carcinoma; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All cohorts (Experimental): NG-350A and pembrolizumab
  Interventions: Biological: NG-350A plus Pembrolizumab

INTERVENTIONS:
Biological: NG-350A plus Pembrolizumab — Patients receive three doses of NG-350A by intravenous infusion and a single dose of Pembrolizumab by intravenous infusion
  Other Names: KEYTRUDA®

SUMMARY:
This is a phase 1a/1b, multicentre, open-label, non-randomized study of NG-350A in combination with pembrolizumab in patients with metastatic or advanced epithelial tumours.

DETAILED DESCRIPTION:
Phase 1a will investigate NG-350A administration by intravenous (IV) infusion in combination with fixed-dose pembrolizumab in patients with metastatic or advanced tumours.

Phase 1b will further investigate the efficacy and safety of the selected dose regimen in up to three of the tumour types evaluated in Phase 1a.

ELIGIBILITY:
Inclusion Criteria:

Phase 1a

1. Patients must have histologically or cytologically documented metastatic or advanced epithelial cancer that has relapsed from or is refractory to standard treatment, or for which no standard treatment is available.
2. At least one measurable site of disease according to RECIST v1.1 criteria; this lesion must be either (i) outside a previously irradiated area or (ii) progressive if it is in a previously irradiated area
3. Tumour accessible for biopsy, biopsy deemed safe by the Investigator, and patient willing to consent to tumour biopsies
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

All patients

1. Provide written informed consent to participate
2. Aged 18 years or over on day of signing informed consent
3. Predicted life expectancy of ≥6 months
4. Adequate lung reserve
5. Adequate renal function
6. Adequate hepatic function
7. Adequate bone marrow/haematological function
8. Meeting reproductive status requirements

Exclusion criteria

1. Prior or planned allogeneic or autologous bone marrow or tissue/organ transplantation
2. Splenectomy
3. Active infections requiring systemic anti-infective treatment, physician monitoring/hospital admission or recurrent fevers (>38.0˚C) associated with a clinical diagnosis of active infection
4. Treatment with the antiviral agents: ribavirin, adefovir, lamivudine, cidofovir or paxlovid within 10 days prior to the first dose of study treatment; or pegylated interferon in the 4 weeks before the first dose of study treatment
5. Known history of hepatitis B infection or known active hepatitis C infection. Known history of HIV infection
6. Patients who have active autoimmune disease that has required systemic therapy in the past 2 years, are immunocompromised in the opinion of the Investigator, or are receiving chronic systemic immunosuppressive treatment
7. Treatment with any live, live-attenuated or COVID-19 vaccine in the 30 days before first dose of study drug
8. Treatment with any other vaccine (including known non live/live-attenuated or non-adenoviral COVID-19 vaccines) in the 7 days before first dose of study drug
9. History of prior Grade 3-4 acute kidney injury or other clinically significant renal impairment
10. History of clinically significant interstitial lung disease or non-infectious pneumonitis/interstitial lung disease that required steroids (or current pneumonitis/interstitial lung disease)
11. Lymphangitic carcinomatosis
12. Infectious or inflammatory bowel disease in the 3 months before the first dose of study treatment
13. Any known CTCAE Grade ≥2 coagulation abnormality/coagulopathy
14. Any clinically significant cardiovascular, peripheral vascular, cerebrovascular, or thromboembolic event in the 6 months before the first dose of study treatment
15. Grade 3 or 4 gastrointestinal bleeding (or risk factors for gastrointestinal bleeding), haemoptysis, or any history of bleeding requiring an investigative procedure, transfusion or hospitalization in the 6 months before the first dose of study treatment
16. Tumour location/extent considered by the Investigator to present a significant risk if tumour flare or necrosis were to occur
17. Use of the following prior therapies/treatments :

    * Treatment with any other enadenotucirev-based virus (parent virus or transgene-modified variants), or anti-CD40 antibody at any time
    * Radiation therapy to the lung that is >30Gy within 6 months of the first dose of trial treatment
    * Treatment with an investigational or licensed anti-cancer monoclonal antibody (mAb), immune checkpoint inhibitor, immune stimulatory treatment or other biological therapy in the 28 days prior to the first dose of study treatment.
    * Prior anti-PD-1 / PD-L1 therapy is permitted without a 'washout' phase
    * Treatment with an investigational or licensed chemotherapy, targeted small molecule or other investigational drug in the 14 days or five half-lives (whichever is shorter) before the first dose of study treatment
    * Major surgery in the 28 days before the first dose of study treatment or radiation therapy in the 14 days before the first dose of study treatment
    * Bisphosphonate therapy or treatment with Receptor Activator of Nuclear factor Kappa-Β (RANK)-ligand inhibitors for metastatic bone disease is permitted
18. All toxicities attributed to prior anti-cancer therapy must have resolved to Grade 1 or baseline before the first dose of study treatment. (see protocol for exceptions)
19. Participants with a history of radiation pneumonitis are not eligible for inclusion
20. Discontinuation from prior treatment with an anti-PD-1 or anti PD L1/PD-L2 agent, or an agent directed to another stimulatory or co-inhibitory T cell receptor, due to a Grade ≥3 immune-related AE
21. Known allergy or hypersensitivity (Grade ≥3) to NG-350A transgene, pembrolizumab and/or any of its excipients or other monoclonal antibodies
22. Known hypersensitivity to both cidofovir and valacyclovir
23. Other prior malignancy active within the previous 3 years (see protocol for exceptions)
24. Known active central nervous system metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and have not required steroid treatment for at least 14 days prior to first dose of study treatment
25. Positive pregnancy test prior to treatment (a serum test must be performed within 24 hours)
26. History or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
27. Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (safety and tolerability) | 100 days after last dose of study drug
  Assess the safety and tolerability of NG-350A in combination with pembrolizumab by review of adverse events including serious adverse events, adverse events leading to study treatment or study discontinuation, and adverse events resulting in death.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Providence Medical Foundation, Santa Monica, California
  - UCLA, Santa Monica, California
  - Moffitt-Advent Health Clinical Research Unit, Celebration, Florida
  - Perelman Center of Advanced Medicine, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- United Kingdom (2):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, Lancashire
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire

REFERENCES:
- [Derived] Naing A, Khalil D, Rosen O, Camidge DR, Lillie T, Ji RR, Stacey A, Thomas M, Rosen L. First-in-human clinical outcomes with NG-350A, an anti-CD40 expressing tumor-selective vector designed to remodel immunosuppressive tumor microenvironments. J Immunother Cancer. 2024 Oct 15;12(10):e010016. doi: 10.1136/jitc-2024-010016. PMID 39414325
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458